CLINICAL TRIAL: NCT03470207
Title: The Prospective Risk Factor Evaluation and Discovery In Chronic Thromboembolic Pulmonary Hypertension Study
Brief Title: The Prospective Risk Factor Evaluation & Discovery In CTEPH Study
Acronym: PREDICT PH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mark W. Dodson (Other)
Responsible Party: Sponsor-Investigator, Mark W. Dodson, Medical Director, CTEPH Program, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1050516
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-Intervention Cohort (Aim 1) (No Intervention): This arm will not have the intervention of the implementation of the structured post-pulmonary embolism follow up protocol that is outlined in Aim 1.
- Pre-Intervention Cohort (Aim 3) (Experimental): This arm will have the intervention of the implementation of the structured post-pulmonary embolism follow up protocol that is outlined in Aim 1.
  Interventions: Procedure: Post-pulmonary embolism follow up protocol

INTERVENTIONS:
Procedure: Post-pulmonary embolism follow up protocol — Structured post-pulmonary embolism follow up protocol (outlined in Aim 1)
  Arms: Pre-Intervention Cohort (Aim 3)

SUMMARY:
This research study wants to find markers in the blood that may help to predict a patient's future risk of developing a disease called CTEPH. The study also wants to see if active monitoring for signs and symptoms of CTEPH after a pulmonary embolism (a blood clot in the lungs) can improve the diagnosis of CTEPH.

Patients who enroll in this study will have periodic blood draws and clinic and/or phone follow-up to monitor for signs and symptoms of CTEPH. Patients' medical records will also be reviewed for information related to pulmonary embolisms and/or CTEPH.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is due to non-resolution of pulmonary embolism (PE), and is the most serious long-term sequela of PE. Without treatment, CTEPH leads to progressive right heart failure and death. Fortunately, most cases of CTEPH are potentially curable by a surgical procedure in which the chronic thromboembolic material is removed from the pulmonary arterial tree, and for those who are not surgical candidates a novel medical therapy is now available. Multiple studies have shown, however, that the majority of CTEPH cases go undiagnosed, and thus many symptomatic patients are never offered these potentially beneficial treatments. Because persistent dyspnea affects up to 50% of patients who survive an acute PE, selecting which patients should undergo further invasive testing for CTEPH is a difficult clinical problem. In this study, the investigators propose to prospectively follow a cohort of high-risk patients after acute PE until CTEPH is either diagnosed or excluded, and perform serial collection and banking of biospecimens that will allow for prospective and longitudinal screening of biomarkers that might predict future risk of CTEPH. Biomarker screening will initially be focused on a panel of 20 pre-specified plasma proteins with roles in coagulation/fibrinolysis or inflammation, as well as assays of fibrinolysis, as these are processes that existing literature suggests are linked to the pathophysiology of CTEPH. The biorepository created for this study could also be used in the future to perform unbiased screening with proteomic techniques or RNAseq in the hopes of identifying novel biomarkers and novel biological processes that are relevant to the development of CTEPH. As there is no current consensus as to whether structured follow-up after PE to detect signs and symptoms of CTEPH is beneficial, this study also includes an analysis of whether a novel structured follow-up program improves identification of incident CTEPH cases. This study has the potential to dramatically improve post-PE care by facilitating stratification of patients by future risk of CTEPH at the time of acute PE, thus allowing for expert follow-up to be tailored to those patients at highest risk for CTEPH. The investigators hope that these efforts will improve the rate at which CTEPH cases are identified, so that more patients can benefit from existing treatments.

ELIGIBILITY:
Inclusion Criteria:

i. Age ≥ 18 years.

ii. Presence of pulmonary embolism (PE) objectively diagnosed by ventilation/perfusion (V/Q) scan or computed tomography pulmonary angiography (CTPA).

iii. Plus one of:

* Prior history of PE before the index event (predicted 2-year incidence of chronic thromboembolic pulmonary hypertension (CTEPH) of 35%).
* Transthoracic echocardiogram (TTE) performed within 72 hours of PE diagnosis demonstrating a maximum velocity of the tricuspid regurgitant (TR) jet ≥ 3.0 meters/second (predicted 2-year incidence of CTEPH of approximately 25%).
* CTPA demonstrating involvement of one of the main pulmonary arteries with PE (predicted 2-year incidence of CTEPH of approximately 15%).
* CTEPH prediction score ≥ 6 (this score is based on several clinical factors, including unprovoked nature of the PE, presence of right ventricular dysfunction by CTPA or TTE, presence of hypothyroidism or diabetes, and thrombolytic therapy for PE).

Exclusion Criteria:

i. The patient previously met diagnostic criteria for pulmonary hypertension of any cause.

ii. Presence of significant left ventricular systolic dysfunction (defined by left ventricular ejection fraction ≤ 45% by TTE), or left sided valvular disease (including mitral or aortic regurgitation or stenosis).

iii. Age > 85 years.

iv. The presence of metastatic malignancy (due to the expected limitation of lifespan to less than the study follow-up period of 2 years).

v. The presence of a significant psychiatric disorder or significant cognitive impairment, which would make follow-up and/or symptom reporting difficult.

vi. Inability or unwillingness to attend follow-up clinic appointments at Intermountain Medical Center (including geographical, financial, and insurance limitations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Chronic Thromboembolic Pulmonary Hypertension (CTEPH) diagnosis rate | Day of diagnosis of pulmonary embolism (PE) until 2 years after day of diagnosis of PE
  Number of CTEPH diagnoses divided by number of patients in each cohort (pre- and post-intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Dodson, MD PhD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Per the consent: "The scientific results from this study may be reported at scientific discussions or published in medical journals. You will not be identified personally in any presentation or published report." "If your samples and data are shared with researchers at other hospitals and institutions outside of Intermountain Healthcare, they will be labeled with a de-identified code so that researchers outside of Intermountain Healthcare will not be able to identify you."
Supporting Information: Study Protocol, ICF
Time Frame: Available: After the end of the study For how long: Indefinite
Access Criteria: Appropriate data sharing agreements must be established with Intermountain Healthcare prior to any sharing of individual participant data.